CLINICAL TRIAL: NCT03985267
Title: Efficacy of Mindfulness Based Swinging Technique (MBST) for Improving Anxiety, Stress, Hopelessness and Self Efficacy Among Breast Cancer Patients in Treatment
Brief Title: A New Mindfulness Intervention Called Mindfulness Based Swinging Technique (MBST) for Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Ozan BAHCIVAN, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/14-01
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Anxiety; Stress; Self Efficacy; Depression; Breast Cancer Female; Hopefulness
Keywords: mindfulness; breast cancer; psycho-oncology; clinical health psychology; ontology; swinging effect intervention; breathing technique; guided imagery; cognitive behavioural therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; Breast Neoplasms | interventions — Cognitive Behavioral Therapy; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Swinging Technique (MBST) (Experimental): Standard guided imagery combined with Mindfulness and breathing technique will be applied. Additionally, the directives will be given to participants to imagine themselves swinging in a green peaceful environment where they will face no harm but healing and full of wellness. Every time they imagine their swing goes up, patient will be asked to physically take a deep breath (taking the breath will be physically (actually) done, not imagining), and when going down patient will be asked to physically release their breath (releasing breath will be physically (actually) done, not imagining).
  Interventions: Behavioral: Mindfulness based Swinging Effect Intervention
- Standard Treatment (Active Comparator): Participants will receive a session of standard psycho-social care for anxiety (50 minutes length). The standard psycho-social care interventions involve the most well-known talking therapy approach of Cognitive Behavioural Therapy (CBT).
  Interventions: Behavioral: Mindfulness based Swinging Effect Intervention

INTERVENTIONS:
Behavioral: Mindfulness based Swinging Effect Intervention — Participants will receive psycho-education about mindfulness and how it operates. That will also assist patients to warm up for the actual intervention. Then the actual swinging effect intervention will commence respectively.
  Other Names: Breathing Technique; Guided Imagery Technique; Cognitive Behavioural Therapy (CBT); Mindfulness

SUMMARY:
It is hypothesised to find that the new mindfulness intervention of Mindfulness Based Swinging Technique (MBST) for Women With Breast Cancer is an effective therapeutic intervention to be applied in breast cancer population. This intervention intended to support patients' management of their chronic illness (self-efficacy) by increasing their hope about their treatment and alleviate anxiety, as well as increase patient saturation level. Therefore, enabling patients to continue to their medical as well as psychological treatment will result improved anxiety, stress levels, hope and self-efficacy. It is known that mental health needs of cancer patients differ from people who do not suffer from a chronic illness.

DETAILED DESCRIPTION:
Participation in this research is entirely voluntary. Participants are required to complete a semi-screening assessment form which asks socio-demographic and bio-medical information. This form is also assess participants eligibility to take part. Then will ask participants to complete the Hospital and Depression Scale (HADS), Self-Efficacy for Managing Chronic Disease (SEMCD), Beck's Hopelessness Scale (BHS), Emotion Thermometer (ET), State Trait Anxiety Inventory (STAI) before and after (pre-post) their allocated intervention (arm). Participants have the right to answer as many or as few questions asked as they wish. They also have the right to withdraw from the study up to four weeks after they have completed the required psychometric measurement tools. Should they wish to withdraw then they will need to inform the researcher by email, quoting their unique participation identification code which will be generated before beginning the study using their name initials and date of birth. This will enable researcher to identify all the materials that needs to be deleted due to their withdrawal from the project. Alternatively, if they decide that they no longer want to take part in the study they can notify the researcher/clinician immediately and their recorded information (if any) will be completely erased from the study. Other than answering a number of demographic questions (in order to establish the characteristics of the sample), participants will not be directly disclosing any confidential personal information. However, the survey completion data will be checked for any identifying information and anonymised if necessary. Participants will be allocated a code number, and this will be used when quoting from the data-set. The data will be kept confidential and stored in a safe locked cabinet/storage at all times. The ethical approval is obtained from one of the Turkish institution where they issue ethical approval in accordance with the ethical standards of the Helsinki declaration.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 and over who can consent
2. Only women participants
3. Diagnosed with breast cancer
4. Native Turkish speaker
5. Currently under cancer treatment (not in remission)
6. Score at least 10 points for Hospital and Depression Scale (5 for anxiety, 5 for depression)
7. Score at least 6 points for Self-Efficacy for Managing Chronic Disease (in overall)
8. Score at least 2 points for the Beck's Hopelessness Scale (in overall)
9. Score at least 20 points for State Trait Anxiety Inventory.

Exclusion Criteria:

1. Being illiterate
2. Having any type of psychiatric history
3. Currently being on psychiatric/neurological medication
4. Having mental retardation
5. Having a fear of swings/swinging
6. Having a severe respiratory illness/severe difficulty in breathing
7. Suffering from any asthmatic or epileptic illnesses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only biological gender will be considered
Enrollment: 156 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the immediate efficacy of the Mindfulness Based Swinging Technique (MBST) to reduce stress and anxiety | 20minutes
  To assess the immediate outcome of the Mindfulness Based Swinging Technique (MBST) whether it is an effective and reliable intervention to reduce stress and anxiety for breast cancer patients. To calculate the total State Trait Anxiety Inventory score (range 20 - 80): the positive items (calm, relaxed, content) will be reverse scored so 1=4, 2=3, 3=2 and 4=1; sum all six scores; multiply total score by 20/6; according to Spielberger's manuals a 'normal' score is approx. 34 - 36.
Evaluation of the immediate efficacy of the Mindfulness Based Swinging Technique (MBST) to increase self-efficacy | 20 minutes
  To assess the immediate outcome of the Mindfulness Based Swinging Technique (MBST) whether it is an effective and reliable intervention to increase self-efficacy for breast cancer patients. In order to assess the effectiveness, Self-Efficacy for Managing Chronic Disease (SEMCD) will be used right before and after the intervention. If two consecutive numbers are circled, the lower number will be coded (less self-efficacy). The score for the scale is the mean of the six items. If more than two items will be missing, scoring the scale will not happen. Higher number indicates higher self-efficacy.The higher values represent a better outcome for this scale.
Evaluation of the immediate efficacy of the Mindfulness Based Swinging Technique (MBST) to increase hopefulness | 20 minutes
  To assess the immediate outcome of the Mindfulness Based Swinging Technique (MBST) whether it is an effective and reliable intervention to increase hopefulness for breast cancer patients. In order to assess the effectiveness, Beck's Hopelessness Scale (BHS) will be used right before and after the intervention. The total score ranges from 0 to 20, the scores will be summed up together with higher levels of hopelessness indicated by higher scores on the scale. The higher values represent a better outcome for this scale.
Evaluation of the long lasting efficacy of the Mindfulness Based Swinging Technique (MBST) to increase self-efficacy | 8 weeks
  To assess the long term follow up outcome of the Mindfulness Based Swinging Technique (MBST) whether it is an effective and reliable intervention to increase self-efficacy for breast cancer patients. In order to assess the effectiveness, Self-Efficacy for Managing Chronic Disease (SEMCD) will be used before and after the intervention. Each of the 6 items are rated from 1 (not at all confident) to 10 (totally confident). The overall score is derived from the mean of the 6 items. The total minimum score will be 6 (very low self-efficacy), and maximum total score will be 60 (very high self-efficacy). Higher scores indicate a better self-efficacy.
Evaluation of the long lasting efficacy of the Mindfulness Based Swinging Technique (MBST) to increase hopefulness | 8 weeks
  To assess the long term follow up outcome of the Mindfulness Based Swinging Technique (MBST) whether it is an effective and reliable intervention to increase hopefulness for breast cancer patients. In order to assess the effectiveness, Beck's Hopelessness Scale (BHS) will be used before and after the intervention. The total score ranges from 0 to 20, the scores will be summed up together with higher levels of hopelessness indicated by higher scores on the scale. The higher values represent a better outcome for this scale.
Evaluation of the long lasting efficacy of the Mindfulness Based Swinging Technique (MBST) to reduce stress and anxiety using the State Trait Anxiety Inventory. | 8 weeks
  To assess the long term follow up of the Mindfulness Based Swinging Technique (MBST) for reducing stress and anxiety State Trait Anxiety Inventory will be used before and after the intervention. To calculate the total State Trait Anxiety Inventory score (range 20 - 80): the positive items (calm, relaxed, content) will be reverse scored so 1=4, 2=3, 3=2 and 4=1; sum all six scores; multiply total score by 20/6; according to Spielberger's manuals a 'normal' score is approx. 34 - 36.
Evaluation of the long lasting efficacy of the Mindfulness Based Swinging Technique (MBST) to reduce stress and anxiety using Emotion Thermometer. | 8 weeks
  To assess the long term follow up of the Mindfulness Based Swinging Technique (MBST) for reducing stress and anxiety Emotion Thermometer will be used before and after the intervention. To calculate the Emotion Thermometer the fixed cut-offs will be used meaning that 0-3 (low) and 4-10 (high) on each component.
Evaluation of the long lasting efficacy of the Mindfulness Based Swinging Technique (MBST) to reduce stress and anxiety using the Hospital Anxiety and Depression Scale. | 8 weeks
  To assess the long term follow up of the Mindfulness Based Swinging Technique (MBST) for reducing stress and anxiety Hospital Anxiety and Depression Scale will be used before and after the intervention. To calculate Hospital Anxiety and Depression Scale the cut of scores are 0-7 considered in normal range, 8-10 considered in Borderline abnormal (borderline case) and 11-21 considered in Abnormal (case) respectively.

SECONDARY OUTCOMES:
Impact of education level on efficacy of the Mindfulness Based Swinging Technique (MBST) | 20 minutes to 8 weeks
  To observe whether breast cancer patients' education level has any impact on efficacy of the Mindfulness Based Swinging Technique (MBST) to reduce anxiety and increase self-efficacy and hopefulness. The participants' education level will be obtained from self-reported socio-demographic semi-screening assessment form.
Impact of marital status on efficacy of the Mindfulness Based Swinging Technique (MBST) | 20 minutes to 8 weeks
  To observe whether breast cancer patients' marital status has any impact on efficacy of the Mindfulness Based Swinging Technique (MBST). The participants' marital status will be obtained from self-reported socio-demographic semi-screening assessment form.
Impact of living arrangements on efficacy of the Mindfulness Based Swinging Technique (MBST) | 20 minutes to 8 weeks
  To observe whether breast cancer patients' living arrangement has any impact on efficacy of the Mindfulness Based Swinging Technique (MBST). The participants' living arrangement status will be obtained from self-reported socio-demographic semi-screening assessment form.
Impact of time for learning cancer diagnosis on efficacy of the Mindfulness Based Swinging Technique (MBST) | 20 minutes to 8 weeks
  To observe whether breast cancer patients' time for learning their cancer diagnosis has any impact on efficacy of Mindfulness Based Swinging Technique (MBST). The information of when participants have learnt their cancer diagnosis will be obtained from self-reported socio-demographic semi-screening assessment form.
Impact of having any metastasis on efficacy of the Mindfulness Based Swinging Technique (MBST) | 20 minutes to 8 weeks
  To observe whether breast cancer patients' metastatic status has any impact on efficacy of Mindfulness Based Swinging Technique (MBST). The participants' metastatic status will be obtained from self-reported socio-demographic semi-screening assessment form.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Maldonado, PhD, MSc, Study Director — University of Barcelona
Locations (2):
- Turkey (Türkiye) (2):
  - Ozel Oz Psikoloji Aile Danisma Merkezi (Oz Psychology Family Counselling Centre), Izmir, Konak
  - EgeMed Hospital, Aydin, Soke

IPD SHARING:
Plan to Share IPD: Yes
data results and outcome will be available to researchers once it is published on a journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: within 1 year of completion of the study.
Access Criteria: it is available through international publication below.
  https://doi.org/10.3389/fpsyg.2022.1007065
  https://doi.org/10.3389/fpsyg.2022.863857

REFERENCES:
- [Background] Bahcivan O, Estape T, Gutierrez-Maldonado J. The swinging effect intervention: CBT based guided imagery and breathing technique integrated with mindfulness therapy for cancer patients. Med Hypotheses. 2018 Dec;121:42-43. doi: 10.1016/j.mehy.2018.09.007. Epub 2018 Sep 6. No abstract available. PMID 30396486
- [Result] Bahcivan O, Estape T, Gutierrez-Maldonado J. Efficacy of New Mindfulness-Based Swinging Technique Intervention: A Pilot Randomised Controlled Trial Among Women With Breast Cancer. Front Psychol. 2022 Jul 4;13:863857. doi: 10.3389/fpsyg.2022.863857. eCollection 2022. PMID 35859820
- See also: Related Info — https://doi.org/10.3389/fpsyg.2022.1007065